CLINICAL TRIAL: NCT02669524
Title: Dissection of the Gastrointestinal-mediated Glucose Disposal and Incretin Defect in Patients With Type 2 Diabetes - the Role of Glucagon
Brief Title: Dissection of the Gastrointestinal-mediated Glucose Disposal and Incretin Defect in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Sofie Hædersdal, MD, PhD student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-15007312
Record Dates: First submitted 2015-12-14; First posted 2016-02-01 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant; Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- T2D + OGTT + LY2409021 (Active Comparator): Type 2 diabetes patients + 50 oral glucose tolerance test 4 hours + the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021; Procedure: OGTT
- T2D + OGTT + placebo (Placebo Comparator): Type 2 diabetes patients + 50 oral glucose tolerance test 4 hours + placebo comparator to the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021 placebo; Procedure: OGTT
- T2D + IIGI + LY2409021 (Active Comparator): Type 2 diabetes patients + isoglycaemic iv glucose infusion + the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021; Procedure: IIGI
- T2D + IIGI + placebo (Placebo Comparator): Type 2 diabetes patients + isoglycaemic iv glucose infusion + placebo comparator to the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021 placebo; Procedure: IIGI
- T2D + MEAL + LY2409021 (Active Comparator): Type 2 diabetes patients + Standardised liquid meal + the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021; Procedure: Standardised liquid meal
- T2D + MEAL + placebo (Placebo Comparator): Type 2 diabetes patients + Standardised liquid meal + placebo comparator to the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021 placebo; Procedure: Standardised liquid meal
- CTRL + OGTT + LY2409021 (Active Comparator): Healthy controls + 50 oral glucose tolerance test 4 hours + the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021; Procedure: OGTT
- CTRL + OGTT + placebo (Placebo Comparator): Healthy controls + 50 oral glucose tolerance test 4 hours + placebo comparator of the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021 placebo; Procedure: OGTT
- CTRL + IIGI + LY2409021 (Active Comparator): Healthy controls + isoglycaemic iv glucose infusion + the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021; Procedure: IIGI
- CTRL + IIGI + placebo (Placebo Comparator): Healthy controls + isoglycaemic iv glucose infusion + placebo comparator the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021 placebo; Procedure: IIGI
- CTRL + MEAL + LY2409021 (Active Comparator): Healthy controls + Standardised liquid meal + the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021; Procedure: Standardised liquid meal
- CTRL + MEAL + placebo (Placebo Comparator): Healthy controls + Standardised liquid meal + placebo comparator of the human antagonist of the glucagon receptor.
  Interventions: Drug: LY2409021 placebo; Procedure: Standardised liquid meal

INTERVENTIONS:
Drug: LY2409021
  Arms: CTRL + IIGI + LY2409021; CTRL + MEAL + LY2409021; CTRL + OGTT + LY2409021; T2D + IIGI + LY2409021; T2D + MEAL + LY2409021; T2D + OGTT + LY2409021
Drug: LY2409021 placebo
  Arms: CTRL + IIGI + placebo; CTRL + MEAL + placebo; CTRL + OGTT + placebo; T2D + IIGI + placebo; T2D + MEAL + placebo; T2D + OGTT + placebo
Procedure: OGTT
  Arms: CTRL + OGTT + LY2409021; CTRL + OGTT + placebo; T2D + OGTT + LY2409021; T2D + OGTT + placebo
Procedure: IIGI
  Arms: CTRL + IIGI + LY2409021; CTRL + IIGI + placebo; T2D + IIGI + LY2409021; T2D + IIGI + placebo
Procedure: Standardised liquid meal
  Arms: CTRL + MEAL + LY2409021; CTRL + MEAL + placebo; T2D + MEAL + LY2409021; T2D + MEAL + placebo

SUMMARY:
In patients with type 2 diabetes, the incretin effect is markedly reduced contributing to the relative insulin deficiency that characterizes these patients. This defect is believed to be due to a decreased effect of GLP-1 and an almost ceased effect of GIP. Nevertheless, the impact of the defect on glucose tolerance is not fully understood. The so-called gastrointestinal-mediated glucose disposal (GIGD) is a measure of glucose handling, which includes the incretin effect, but also other factors affecting glucose disposal (e.g. glucagon secretion). Interestingly, patients with type 2 diabetes exhibit elevated plasma glucagon levels in the fasting state, and glucagon concentrations fail to decrease appropriately and may even increase in response to ingestion of glucose and show exaggerated increases after a mixed meal. With the current project the investigators wish to elucidate how this paradoxical glucagon response observed in patients with type 2 diabetes affects the GIGD, the incretin effect and postprandial glucose excursions.

Ten patients with type 2 diabetes and 10 healthy matched control subjects will be enrolled in this randomised, placebo-controlled, double-blinded study. The aim is to examine the effect of a glucagon receptor antagonist (GRA) on gastrointestinal-mediated glucose disposal (GIGD), incretin effect and postprandial glucose excursions in patients with type 2 diabetes and healthy controls. Participants will attend two oral glucose tolerance tests (OGTT), two isoglycaemic iv glucose infusion (IIGI) and two standardised liquid meals.

ELIGIBILITY:
Inclusion Criteria:

Patients with type 2 diabetes

* Caucasians above 35 years of age with diet or metformin treated type 2 diabetes for at least 3 month (diagnosed according to the criteria of the World Health Organization (WHO)
* Normal haemoglobin
* Informed consent

Healthy subjects

* Normal fasting plasma glucose (FPG) <6.1 mmol/l and HbA1c <42 mmol/mol (6.0%)
* Normal haemoglobin
* Age above 35 years
* Informed consent

Exclusion Criteria:

Patients with type 2 diabetes

* Inflammatory bowel disease
* Intestinal resections
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2×normal values)
* Treatment with medicine that cannot be paused for 12 hours
* Pregnancy and/or breastfeeding
* Family history of pancreatic islet tumours
* Age above 80 years

Healthy subjects

* Diabetes or prediabetes with reduced glucose tolerance: FPG >6.0 mmol/l and/or HbA1c >42 mmol/mol
* First degree relatives with type 2 diabetes
* Inflammatory bowel disease
* Intestinal resections
* Treatment with medicine that cannot be paused for 12 hours
* Pregnancy and/or breastfeeding
* Age above 80 years

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Differences in GIGD (%) | Comparison between experimental days with and without the glucagon receptor antagonist . The glucose disposal at time 240 minutes will be used.
  GIGD = Gastrointestinal glucose disposal. GIGD (%) = 100% × (glucoseOGTT-glucoseIIGI)/glucoseOGTT.
Difference in postprandial glucose excursions | Area under the curve (AUC) time frame: 0, 5, 10, 15, 20, 25, 30, 40, 50, 60, 70, 80, 90, 105, 120, 150, 180, 210, 240 minutes. Comparison between experimental days with and without the glucagon receptor antagonist.
  Difference in postprandial glucose excursions (measured as incremental (baseline substracted) area under the curve (AUC) values).

SECONDARY OUTCOMES:
Incretin effect | Insulin AUC time frame: 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes. Comparison between experimental days with and without the glucagon receptor antagonist
  The incretin effect (100% × [β-cell secretory response to oral glucose tolerance test - intravenous β-cell secretory response]/β-cell secretory response to oral glucose tolerance test)
Endogenous glucose production | Plasma concentration of 6,6^2 H2-glucose and U-13C^6-glucose at times: 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes.
  Glucose rate of appearance will be calculated by the non-steady state equation using double tracer technique.
Lipolysis | Plasma concentration of 1,1,2,3,3-^2-H5 - glycerol measured at times: 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes.
  Glycerol disappearance will be calculated by the non-steady state equation using double tracer technique.
Serum/plasma concentrations of insulin, C-peptide, glucagon, GIP and GLP-1. | Time frame: 0,10, 20, 30, 50, 60, 70, 90, 105, 120, 150, 240 minutes.
  Insulin, C-peptide, glucagon, GIP and GLP-1 serum/plasma concentrations will be measured in pM.
Appetite | VAS scales will be handed out at time 0, 30, 60, 90, 120, 150, 180 and 240 minutes.
  Appetite will be evaluated with a visual analogue scale (VAS).
Energy intake (kcal/kJ) | At time 240 to 270, the participants will eat an ad libitum meal. Comparison between experimental days with and without the glucagon receptor antagonist
  At the end of the clamp experiment food intake will be examined with an ad libitum meal. The weight of the food will be measured i grams and calculated to the energy intake in kcal/kJ.
Changes in blood pressure (mmHg) | Measured at time 0 and time 210 minutes. Comparison between experimental days with and without the glucagon receptor antagonist
Changes in pulse rate (beat per minute) | Measured at time 0 and at time 210 minutes. Comparison between experimental days with and without the glucagon receptor antagonist
Differences in gastric emptying | -30,-15, 0, 10, 20, 30, 50, 70, 90, 105, 120, 150, 240 minutes
  Measurement of p-paracetamol. Measurement of time to peak and incremental area under the curve (iAUC)
Free fatty acids | -30,-15, 0, 10, 20, 30, 50, 70, 90, 105, 120, 150, 240 minutes
  serum values of free fatty acids
Fibroblast growth factor-21 | -30,-15, 0, 10, 20, 30, 50, 70, 90, 105, 120, 150, 240 minutes
  plasma values of FGF-21

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Copenhagen University, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided